CLINICAL TRIAL: NCT02062541
Title: Effect of Functional Assessment and Immediate Rehabilitation of ED Admitted Elderly With Reduced Functional Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Sygehus Lillebaelt (Other)
Responsible Party: Principal Investigator, Christian Backer Mogensen, associate professor, University of Southern Denmark
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: SLB-ED-02-2014
Record Dates: First submitted 2014-02-12; First posted 2014-02-13 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Functionally-Impaired Elderly
Keywords: functional assessment; rehabilitation; cross-sectorial cooperation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Funct. assessment+fast rehabilitation (Experimental): Funct. assessment+fast rehabilitation
  Interventions: Other: Funct. assessment+fast rehabilitation
- Funct. assessment+usual rehabilitation (Experimental): Funct. assessment+usual rehabilitation
  Interventions: Other: Funct. assessment+usual rehabilitation
- usual assessment+fast rehabilitation (Experimental): usual assessment+fast rehabilitation
  Interventions: Other: usual assessment+fast rehabilitation
- usual assessment+usual rehabilitation (No Intervention): usual assessment+usual rehabilitation

INTERVENTIONS:
Other: Funct. assessment+fast rehabilitation
  Arms: Funct. assessment+fast rehabilitation
Other: Funct. assessment+usual rehabilitation
  Arms: Funct. assessment+usual rehabilitation
Other: usual assessment+fast rehabilitation
  Arms: usual assessment+fast rehabilitation

SUMMARY:
Background: Illness and hospitalisation, even of short duration, pose separate risks for permanently reduced functional performance in elderly medical patients. Functional assessment in the acute pathway will ensure early detection of declining performance and form the basis for mobilisation during hospitalisation and subsequent rehabilitation. For optimal results rehabilitation should begin immediately after discharge.

The aim of this study is to investigate the effect of a systematic functional assessment in the emergency departments (ED) of elderly medical patients with reduced functional performance when combined with immediate post-discharge rehabilitation.

Method/design: The study is a two-way factorial randomised clinical trial. Participants will be recruited among patients admitted to the ED who are above 65 years of age with reduced functional performance. Patients will be randomly assigned to one of four groups: 1) functional assessment and immediate rehabilitation; 2) functional assessment and usual rehabilitation; 3) usual assessment and immediate rehabilitation; 4) usual assessment and usual rehabilitation.

Primary outcome: 30-second chair-stand test administered at admission and two weeks after discharge.

We hypothesise that such assessment in the ED or/and immediate rehabilitation will result in sustained or improved performance in comparison to regimen in which neither of these interventions are offered.

ELIGIBILITY:
Inclusion Criteria:

* medical patients of 65 years of age or older admitted to the ED
* Can speak and understand Danish
* Resident in either of the two included municipalities
* Can report personal data and decide on consent
* Are able to sit on an chair and perform ≤ 9 repetitions at the 30-s. chair-stand test

Exclusion Criteria:

* Patients suffering from a progressive neurological or cognitive deficit or disease.
* Patients ordinarily unable to walk

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 336 (Actual)
Dates: Start 2015-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
30-second-chair-stand test | up to 14 days after admission date

CONTACTS AND LOCATIONS:
Overall Officials: Christian B Mogensen, PhD, Principal Investigator — University of Southern Denmark
Locations (1):
- Lillebaelt hospital, Kolding, Denmark

REFERENCES:
- [Derived] Bruun IH, Norgaard B, Maribo T, Schiottz-Christensen B, Mogensen CB. The effect on physical performance of a functional assessment and immediate rehabilitation of acutely admitted elderly patients with reduced functional performance: the design of a randomised clinical trial. BMJ Open. 2014 Jun 17;4(6):e005252. doi: 10.1136/bmjopen-2014-005252. PMID 24939812